CLINICAL TRIAL: NCT03021915
Title: Single Center, Prospective Controlled Pilot Study of the OvaPrime Procedure
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: OvaScience, Inc. is no longer study sponsor as it is undergoing a merger. Follow-up will be conducted by sponsor-investigator Dr. Bob Casper.
Sponsor: OvaScience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-P01
Record Dates: First submitted 2016-11-20; First posted 2017-01-16 (Estimated); Last update posted 2018-11-28 (Actual); Status verified 2018-11

CONDITIONS: Primary Ovarian Insufficiency; Poor Ovarian Response
MeSH Terms: conditions — Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OvaPrime Treatment (Other): The treatment is based on identified EggPC cells in the outer-most layer of the ovary. During OvaPrime, the EggPC cells are isolated from biopsy tissue obtained from the outer layer of the ovary. OvaScience separates the EggPC cells and these isolated cells are then returned to the IVF clinic - there is no culture or expansion of the EggPC cells during this process. Upon receipt of the autologous EggPC cells, the clinic initiates the process of reintroducing the cells into the follicular development zone of the woman's own ovary using a laparoscopic procedure. Once in the ovary, the EggPC cells have the opportunity to develop and mature into fertilizable eggs naturally or with controlled ovarian hyperstimulation (when stimulated by exogenous gonadotropins) using standard IVF protocols.
  Interventions: Other: OvaPrime Treatment

INTERVENTIONS:
Other: OvaPrime Treatment — The treatment is based on identified EggPC cells in the outer-most layer of the ovary. During OvaPrime, the EggPC cells are isolated from biopsy tissue obtained from the outer layer of the ovary. OvaScience separates the EggPC cells and these isolated cells are then returned to the IVF clinic - there is no culture or expansion of the EggPC cells during this process. Upon receipt of the autologous EggPC cells, the clinic initiates the process of reintroducing the cells into the follicular development zone of the woman's own ovary using a laparoscopic procedure. Once in the ovary, the EggPC cells have the opportunity to develop and mature into fertilizable eggs naturally or with controlled ovarian hyperstimulation (when stimulated by exogenous gonadotropins) using standard IVF protocols.

SUMMARY:
This is a single center, prospective, controlled pilot safety research study. The primary objective of this research study is to assess the safety with the use of the OvaPrime procedure in women who are diagnosed with either primary ovarian insufficiency (POI) or poor ovarian response (POR).

A maximum of ninety-five (95) subjects will be enrolled consisting of a minimum of thirty (30) POI subjects and a minimum of fifty (50) POR to achieve the target sample size of 70 Modified Intent-to-Treat (mITT) subjects as the primary analysis population. Each subject shall have one ovary exposed to the EggPC cells while the contralateral ovary is exposed to the EggPC vehicle as a means to have each subject serve as their own control. Results between the treatment and control ovary will be examined for relevant endpoints such as antral follicle counts.

The duration of the research study is estimated at approximately 6 years total, for the period spanning enrollment (estimated at approximately six months), eight months to the last hyperstimulation and through completion of 5-year follow-up (main study protocol with one year primary endpoint and LTFU sub-study which extends to 5 additional years).

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who are diagnosed with EITHER POI or POR as defined below:

   * POI subjects who are:

     * < 40 years of age
     * have non-detectable AMH
     * FSH >15.0 mIU/ml and/or symptoms of menopause
   * POR (based on European Society of Human Reproduction and Embryology (ESHRE) guidelines must have two of the following:

     * 40 years of age

       * A previous IVF cycle with < 3 oocytes with a standard of care controlled ovarian hyperstimulation protocol
       * An abnormal ovarian reserve test defined as:

         1. AFC < 5 - 7 follicles or
         2. AMH < 0.5 - 1.1 ng/ml or
         3. Highest ever baseline FSH > 15.0 ml U/ml
2. Subject must have both ovaries.
3. Subject agrees to participate in main study follow up as well as Long Term Follow-up (LTFU) sub-study
4. Subject's male partner or sperm donor source must meet the following requirements:

   * Semen must be an ejaculate (not surgically derived, epididymal, testicular, electro- ejaculated sperm), collected by ejaculation.
   * Male partner's testes must not have been exposed to chemotherapy.
   * Semen must have some morphologically normal spermatozoa according to the World Health Organization (see table below) and adequate concentration with some motile spermatozoa for insemination of all oocytes by intra-cytoplasmic sperm injection (ICSI).

   WHO Semen variable 2010 Volume (mL) 1.5 Concentration (106 mL-1) 15 Total sperm number (106/ejaculate) 39 Motility (% motile) 40 (a + b + c) Forward progression 32 (a + b) Morphology (% normal) 4 Viability/vitality (% live) 58 White blood cells (106 mL-1) < 1.0
5. Partner must also agree to all research study requirements including follow up (including main study as well as LTFU sub-study) of offspring and sign consent form (not applicable in the case of a woman using sperm donation).

Exclusion Criteria:

1. Subject with a diagnosis of POI who is ≥ 40 years of age or < 21 years of age at the time of the OvaPrime procedure
2. Subject with onset of POI < 18 years of age
3. Subject with a diagnosis of POR who is > 45 years of age at the time of the OvaPrime procedure
4. Subject has had any prior surgery/medical condition that would prevent direct access to the ovaries (e.g., pelvic adhesions, tubo- ovarian adhesions location/displacement of the ovary(ies) or high body mass index (BMI)).
5. Subject has severe (stage IV) endometriosis or presence of an endometrioma
6. Subject has a unilateral or bilateral untreated hydrosalpinx
7. Subject has participated in the active phase of another investigational trial within the previous 30 days
8. Subject has a history of prior chemotherapy or radiation therapy to the pelvis
9. Subjects and/or partner (supplying sperm) with known karyotypic abnormalities 10. Subjects with POI who have FMR1 premutations or an FMRI mutation

11. Subjects who are positive for the hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) and human immunodeficiency virus (HIV).

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2016-10; Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Safety - to evaluate the frequency of adverse events (AE) and serious adverse events (SAE) of all subjects regardless of pregnancy. | 2 years
  For subjects who fail to achieve pregnancy, they will be assessed for one year from the date of the OvaPrime procedure. For subjects who become pregnant, they will be followed through the pregnancy and 1-year post-partum. The safety of the off-spring will be monitored by this research study up to one-year post delivery in the main study and for up to 5 years in the long-term follow-up study.

SECONDARY OUTCOMES:
Hormone level change from baseline in the following: anti-mullerian hormone level (AMH), follicle stimulating hormone (FSH) and estradiol (E2) | 1 year
Development of new primordial or growing follicles in the treated ovary as determined by decreasing serum FSH | 1 year
Development of new primordial or growing follicles in the treated ovary as determined by increasing serum AMH | 1 year
Development of new primordial or growing follicles in the treated ovary as determined by the presence of new basal antral follicles on ultrasound | 1 year
Development of new primordial or growing follicles in the treated ovary as determined by increasing serum E2 | 1 year
Egg maturation and developmental potential as evidenced by: Number of MII eggs as assessed by embryologist. | 1 year
Egg maturation and developmental potential as evidenced by: Number of embryos on Day 5 that are graded 3BB or greater as assessed by embryologist | 1 year
Egg maturation and developmental potential as evidenced by: Number of embryo transfers | 1 year
Pre-implantation Genetic Screening (PGS) results | 1 year
The occurrence of pregnancy | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Dan Nayot, MD, Principal Investigator — TRIO Fertility Clinic
Locations (1):
- TRIO, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No